CLINICAL TRIAL: NCT07054957
Title: Use of Handheld Fans in Management of Hot Flashes in Women With Breast Cancer Receiving Hormonetherapy
Acronym: Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Aslıhan ÖZTÜRK ÇETİN, Principal Investigator, Izmir Bakircay University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: Bakırçay Üniversitesi
Record Dates: First submitted 2025-06-03; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Handheld Fan; Hot Flashes; Hormonetherapy
Keywords: breast cancer; hormonetherapy; handheld fan; hot flashes; symptom management
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study was conducted in a single-blind, single-center, randomized controlled design in breast cancer patients receiving hormone therapy in an outpatient chemotherapy unit.
  This study was conducted in the outpatient chemotherapy unit of a training and research university hospital in Turkey between November 2023 and October 2024.: This randomised controlled study was a pretest-posttest experimental design. The study sample consisted of 64 breast cancer patients (n = 32 for each of the intervention and control groups) receiving hormone therapy treatment in the medical oncology department of a university hospital. The intervention group used a hand-held fan when experiencing hot flush symptoms, while the control group did not receive any intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): pre-test, mid-test and final test will be administered.
- İntervention group (Experimental): Group using hand fans
  Interventions: Other: Handheld fan; Other: Control Group

INTERVENTIONS:
Other: Handheld fan — Group using hand fans
  Arms: İntervention group
Other: Control Group — pre-test, mid-test and post-test will be administered.
  Arms: İntervention group

SUMMARY:
Hot flushes are a common symptom in women with breast cancer receiving hormone therapy. It can lead to conditions that reduce quality of life such as sleep quality deterioration, sexual problems and discomfort in daily life. Effective management of the symptom improves the quality of life of patients.

The aim of the study was to examine the effect of handheld fan use in the management of hot flashes in women with breast cancer receiving hormone therapy.

Hypotheses of the research:

H1: Handheld fan use has no effect in managing hot flashes in women with breast cancer receiving hormone therapy. H2: The use of handheld fan has an effect on the management of hot flashes in women with breast cancer receiving hormone therapy. This randomised controlled study was a pretest-posttest experimental design. The study sample consisted of 64 breast cancer patients (n = 32 for each of the intervention and control groups) receiving hormone therapy treatment in the medical oncology department of a university hospital. The intervention group used a hand-held fan when experiencing hot flush symptoms, while the control group did not receive any intervention. The pre-test and post-test Visual Analogue Scale (VAS) and hot flush belief scale scores and the results of the individual identifying information form were compared for both groups.

DETAILED DESCRIPTION:
Study Design This study was conducted in a single-blind, single-center, randomized controlled design in breast cancer patients receiving hormone therapy in an outpatient chemotherapy unit.

This study was conducted in the outpatient chemotherapy unit of a training and research university hospital in Turkey Participants Power analysis was performed to determine the sample size of the study and the power of the test was calculated with G*Power 3.1 programme. Accordingly, with a margin of error of α=.05 and 80% power level, a total of 52 people, 26 people in each group, were found sufficient. This number was increased by 20% in case there were patients who wanted to leave the study. Patients were assigned to the control (n=32) and intervention groups (n=32) by simple randomisation.

The inclusion criteria were patients aged 18 years and over, diagnosed with breast cancer, receiving active hormone therapy, experiencing hot flush symptoms and volunteering to participate in the study. Patients who were in menopause and had verbal and auditory communication problems were excluded from the study.

Randomisation A total of 90 patients who met the inclusion criteria were reached. Since 10 of the 90 patients did not meet the inclusion criteria, 80 patients were assigned to the groups by simple randomisation (40 in the intervention group and 40 in the control group). In order to minimise selection bias, a table of random numbers from the simple random sampling method, which is one of the probability sampling methods, was used. Since 5 of the 40 patients randomly assigned to the intervention group refused to participate in the study and 3 of them continued to receive treatment in another hospital, the study was terminated with 32 patients. Of the 40 patients randomly assigned to the control group, the study was terminated with a total of 32 patients because 6 refused to participate in the study and 2 left due to interruption of treatment.

Measurements Research data were collected using the "Individual Information Form", "Visual Analog Scale (VAS)" and "Hot Flash Belief Scale" prepared by the researchers in line with the literature. Individual Information Form; the form prepared by the researchers consisted of 13 questions regarding the individuals' age, gender, place of residence, number of children, marital status, educational status, employment status, economic status, chronic disease status, duration of cancer diagnosis, cancer stage, treatments received, and practices performed to prevent symptoms15.

Visual Analog Scale (VAS); VAS is used to quantify some values that cannot be measured numerically. It consists of a 10 cm long line at one end, which is expressed as very good for the individual/patient and very bad at the other end. VAS is also a valid and reliable measurement tool for measuring other subjective emotions such as mood. In this study, VAS is preferred for the hot flashes experienced by women with breast cancer receiving hormone therapy.

Hot Flashes Belief Scale; The scale consists of 27 items and three sub-dimensions. The beliefs about oneself in a social context sub-dimension: It was formed with 13 items (1, 6-11, 13,14, 17, 20, 21, 23) that describe how women feel when they experience hot flashes in social environments. The beliefs about coping with hot flashes sub-dimension: It was formed with 10 items (2, 5, 12, 15, 16, 18, 19, 24, 26, 27) that describe beliefs about coping with hot flashes. Beliefs about coping with night sweats sub-dimension: It consists of 4 items (3, 4, 22, 25) describing women's beliefs about coping with night sweats. Each item of the scale is rated on a 6- point Likert type scale ranging from "strongly disagree" (0 points) to "strongly agree" (5 points). It is stated that items 2, 4, 5, 11, 15, 18, 25 of the scale are reverse coded. The total score of the scale varies between 0-135, and a high score on the scale indicates a high level of negative belief. The reliability analysis conducted for the Hot Flash Belief Scale and its sub-dimensions shows that there is a high internal consistency in the scale. The total Cronbach's Alpha value of the scale was calculated as 0.950, and 0.941 for social belief, 0.933 for coping, and 0.946 for night sweats were found for the sub-dimensions. All Alpha values above 0.90 indicate that the scale is a reliable measurement tool in general and at the sub-dimensions.

Data Collection The data of the study were collected by the researcher using face-to-face interview method in the outpatient chemotherapy unit between November 2023 and October 2024. The data collection process took approximately 15-20 minutes. After the patients who met the inclusion criteria were informed about the purpose of the study, the application and the data collection process, their verbal and written consents were obtained. The experimental group (hand fan) who accepted the study were administered the pre-test (Hot flush VAS-Hot Flush Belief Scale) on the first day they came to the outpatient clinic and the post- test (Hot flush VAS-Hot Flush Belief Scale) when they came to the second control (at least 3 months).

Patients in the experimental group were given a hand fan and asked to use the hand fan when they felt hot flushes. They were also reminded to use the hand fan by calling twice a week.

The control group who accepted the study will be administered the pre-test (Hot flush VAS-Hot Flush Belief Scale) on the first day of their visit to the outpatient clinic and the post-test (Hot flush VAS-Hot Flush Belief Scale) on the second visit (at least 3 months).

Data Analysis Data were analyzed using Statistical Social Sciences Package 26.0. Descriptive statistics including mean, standard deviation, frequency, minimum and maximum values were used to evaluate the data. Homogeneity of the study groups was tested using Pearson chi-square analysis and independent samples t-tests. Comparisons of two independent groups were performed using Mann-Whitney U tests and p<.05 was considered statistically significant. Post-hoc power analysis was performed using G*Power software to evaluate the statistical power of ANOVA test in this study. For the analysis, the effect size (f) was determined as 0.25, α error probability was 0.05 and a total sample size of 386 was considered; four groups were considered. The results show that the noncentrality parameter was 24.13, the critical F value was 2.63 and the power (1 - β error probability) value was 99%. These findings reveal that the study has high statistical power and increase the reliability of the results.

Ethical Consideration Prior to the study, approval was obtained from the Izmir Bakırçay University Non-Interventional Clinical Research Ethics Committee (decision no/date: 1266/01.11.2023). The Declaration ofHelsinki was followed at all stages of the study. Informed consent was obtained from all participants and they were given a commitment to withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinical breast cancer
* Experiencing hot flashes

Exclusion Criteria:

- Menopausal women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — MANAGEMENT OF HOT FLASHES IN WOMEN WITH BREAST CANCER RECEIVING HORMONETHERAPY
Enrollment: 64 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Individual Information Form | 12 weeks
  This form contains questions about sociodemographic characteristics, diseases and symptoms.
Visual Analog Scale (VAS) | 12 weeks
  Visual Analog Scale (VAS); VAS is used to quantify some values that cannot be measured numerically. It consists of a 10 cm long line at one end, which is expressed as very good for the individual/patient and very bad at the other end. VAS is also a valid and reliable measurement tool for measuring other subjective emotions such as mood. In this study, VAS is preferred for the hot flashes experienced by women with breast cancer receiving hormone therapy
Hot Flashes Belief Scale | 12 weeks
  The scale consists of 27 items and three sub-dimensions. The beliefs about oneself in a social context sub-dimension: It was formed with 13 items (1, 6-11, 13, 14, 17, 20, 21, 23) that describe how women feel when they experience hot flashes in social environments. The beliefs about coping with hot flashes sub-dimension: It was formed with 10 items (2, 5, 12, 15, 16, 18, 19, 24, 26, 27) that describe beliefs about coping with hot flashes. Beliefs about coping with night sweats sub-dimension: It consists of 4 items (3, 4, 22, 25) describing women's beliefs about coping with night sweats. Each item of the scale is rated on a 6-point Likert type scale ranging from "strongly disagree" (0 points) to "strongly agree" (5 points). It is stated that items 2, 4, 5, 11, 15, 18, 25 of the scale are reverse coded. The total score of the scale varies between 0-135, and a high score on the scale indicates a high level of negative belief.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Bakircay University, Izmir, Seyrek/Menemen, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No